CLINICAL TRIAL: NCT03035201
Title: COcoa Supplement and Multivitamin Outcomes Study-Mind
Brief Title: COcoa Supplement and Multivitamin Outcomes Study for the Mind
Acronym: COSMOS-Mind
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00037753; 1R01AG050657-01A1 (NIH)
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Impairment; Dementia; Aging
Keywords: Memory; Mild Cognitive Impairment; Alzheimer's Disease; Cognition
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cocoa extract + multivitamin (MTV): 2 capsules containing 500 mg/d cocoa extract; daily MTV
- Cocoa extract + multivitamin placebo: 2 capsules containing 500 mg/d cocoa extract; daily MTV placebo
- Cocoa extract placebo + multivitamin: Cocoa extract placebo (2 capsules/d); daily MTV
- Cocoa extract placebo + multivitamin placebo: Cocoa extract placebo (2 capsules/d); daily MTV placebo

SUMMARY:
The parent trial (COcoa Supplement and Multivitamin Outcomes Study, COSMOS; NCT02422745) is a randomized clinical trial of cocoa extract supplement (containing a total of 500 mg/d flavanols, including 80 mg. (-)-epicatechins), and a standard multivitamin supplement to reduce the risk of cardiovascular disease and cancer among men aged 60 years and older and women aged 65 years and older. A cognitive ancillary study (COSMOS-Mind) is being conducted among men and women, 65 years and older, who are enrolled in COSMOS and will examine whether the cocoa extract supplement or the multivitamin supplement improves cognitive function and reduces risk of cognitive impairment, including Alzheimer's disease (AD) and other related types of dementia. Participants at the Wake Forest site will only be getting a phone call.

DETAILED DESCRIPTION:
Identifying a safe, affordable, and well-tolerated intervention that prevents cognitive decline in older adults is of critical public health importance. There is compelling evidence from basic science, and small clinical studies that cocoa flavanols may protect cognitive function in older adults and reduce risk of Alzheimer's disease (AD) and related dementia. Thus, this intervention could have important downstream benefits for health care utilization and cost, caregiver burden, and overall quality of life for older adults. Cocoa flavanol effects on cognition, however, need to be assessed in a definitive clinical trial.

The parent trial (COSMOS) will enroll 21,442 women and men nationwide, drawn from the Women's Health Initiative (WHI) participant cohort and the VITamin D and OmegA-3 TriaL (VITAL) non-randomized respondent cohort, and will be conducted primarily by mail to assess whether high-potency cocoa flavanol extract and a multivitamin - alone or in combination - will reduce risk of cardiovascular disease and cancer over 3 years of follow-up.

After the COSMOS trial began, an advanced method to analyze cocoa flavanols was accredited by Association of Official Agricultural Chemists (AOAC) International as a First Action Official Method of Analysis https://doi.org/10.1093/jaoacint/qsaa132 [secure-web.cisco.com]). This updated method relies on a reference material (RM8403) recently standardized and made commercially available by the U.S. National Institute of Standards and Technology. While the actual cocoa flavanol content of the COSMOS intervention remained unchanged throughout the trial, the application of this new analytical method led to expected changes in how the total cocoa flavanol content is now reported. Applying AOAC 2020.05/RM8403 to the COSMOS intervention, the total cocoa flavanol content of the COSMOS intervention is now 500 mg/day. Reporting of (-)-epicatechin content remained unaffected. Going forward, this record will therefore apply AOAC 2020.05/RM8403 and report that the COSMOS intervention tested 500 mg/day of cocoa flavanols, including 80 mg of (-)-epicatechin.

Once participants are enrolled in COSMOS, the study team at Brigham and Women's Hospital will provide contact information and other parent trial outcomes for COSMOS-Mind participants to the Wake Forest team using a secure web-based data transfer system. This seamless exchange of information between sites will permit timely accounting to ensure that the targeted demographics for enrollment are achieved (e.g. gender, age, race, ethnicity).

COSMOS-Mind will only be administered a telephone cognitive assessment to all participants at enrollment (baseline), and annually for 3 years of follow-up by trained and certified staff of the Wake Forest COSMOS-Mind team.

ELIGIBILITY:
Participants in COSMOS (NCT02422745) who meet the following criteria are eligible to participate in this ancillary study:

Inclusion Criteria -

1. Men and women 65 years and older.
2. Willingness to participate.
3. Ability to answer questions by phone.

Exclusion Criteria -

1. Participants who are co-enrolled in the WHI Memory Study.
2. Participants with insulin-dependent diabetes.
3. Participants who are unable to complete the baseline cognitive assessments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: COSMOS-Mind will include 2,000 participants from the COSMOS parent trial who are at least 65 years of age, with approximately equal distribution of women and men.
Sampling Method: Non-Probability Sample
Enrollment: 2262 (Actual)
Dates: Start 2016-09; Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Baker, PhD, Principal Investigator — Wake Forest University Health Sciences; Mark A Espeland, PhD, Principal Investigator — Wake Forest University Health Sciences; Stephen R Rapp, PhD, Principal Investigator — Co-Investigator Wake Forest School of Medicine; Sally A Shumaker, PhD, Principal Investigator — Co-Investigator Wake Forest School of Medicine; JoAnn E Manson, MD, Principal Investigator — Parent Study Principal Investigator/COSMOS Mind Co-Investigator Brigham and Women's Hospital; Howard Sesso, SCD, MPH, Principal Investigator — Parent Study Principal Investigator/COSMOS Mind Co-Investigator Brigham and Women's Hospital
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
COSMOS-Mind and COSMOS (parent trial, PI: Manson and Sesso) have data transfer procedures and protocols in place which use password protection and encryption, to permit seamless and secure exchange of information. Safety monitoring will be completed through the parent trial. The COSMOS-Mind staff will send all adverse events reported to them to the parent trial for reporting and follow-up. This data will be sent electronically only to approved users through a protected network.
Supporting Information: Study Protocol, ICF
Time Frame: after completion of study
Access Criteria: Data have been submitted to the parent COSMOS trial for merging with phenotypes and distribution.

REFERENCES:
- [Derived] Vyas CM, Manson JE, Sesso HD, Cook NR, Rist PM, Weinberg A, Moorthy MV, Baker LD, Espeland MA, Yeung LK, Brickman AM, Okereke OI. Effect of multivitamin-mineral supplementation versus placebo on cognitive function: results from the clinic subcohort of the COcoa Supplement and Multivitamin Outcomes Study (COSMOS) randomized clinical trial and meta-analysis of 3 cognitive studies within COSMOS. Am J Clin Nutr. 2024 Mar;119(3):692-701. doi: 10.1016/j.ajcnut.2023.12.011. Epub 2024 Jan 18. PMID 38244989
- [Derived] Baker LD, Rapp SR, Shumaker SA, Manson JE, Sesso HD, Gaussoin SA, Harris D, Caudle B, Pleasants D, Espeland MA; COSMOS-Mind Research Group. Design and baseline characteristics of the cocoa supplement and multivitamin outcomes study for the Mind: COSMOS-Mind. Contemp Clin Trials. 2019 Aug;83:57-63. doi: 10.1016/j.cct.2019.06.019. Epub 2019 Jul 2. PMID 31271875
- See also: COcoa Supplement and Multivitamin Outcomes Study — http://www.cosmostrial.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cocoa Extract + Multivitamin: Daily cocoa extract (capsule containing 750 mg/d flavanols, including 75 mg (-)-epicatechin, and 90 mg theobromine) Daily Centrum Silver
- Cocoa Extract + Multivitamin Placebo: Daily cocoa extract (capsule containing 750 mg/d flavanols, including 75 mg (-)-epicatechin, and 90 mg theobromine) Daily Centrum Silver placebo
- Cocoa Extract Placebo + Multivitamin: Daily cocoa extract placebo Daily Centrum Silver
- Cocoa Extract Placebo + Multivitamin Placebo: Daily cocoa extract placebo Daily Centrum Silver placebo
Period: Overall Study
Arm/Group | Cocoa Extract + Multivitamin | Cocoa Extract + Multivitamin Placebo | Cocoa Extract Placebo + Multivitamin | Cocoa Extract Placebo + Multivitamin Placebo
Started | 571 | 553 | 551 | 587
Completed | 444 | 441 | 441 | 462
Not Completed | 127 | 112 | 110 | 125
Not completed — Death | 9 | 12 | 9 | 10
Not completed — Withdrawal by Subject | 51 | 49 | 37 | 46
Not completed — Lost to Follow-up | 67 | 51 | 64 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cocoa Extract + Multivitamin | Cocoa Extract + Multivitamin Placebo | Cocoa Extract Placebo + Multivitamin | Cocoa Extract Placebo + Multivitamin Placebo | Total
Number analyzed (Participants) | 571 | 553 | 551 | 587 | 2262
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (5.5) | 73.2 (5.6) | 72.9 (5.6) | 73.1 (5.7) | 73.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 330 | 319 | 360 | 1348
  Male | 232 | 223 | 232 | 227 | 914
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 2 | 1 | 8 | 2 | 13
  Asian/Pacific Islander | 9 | 12 | 10 | 8 | 39
  Black/African American | 40 | 23 | 34 | 34 | 131
  Hispanic | 13 | 18 | 15 | 21 | 67
  Multiracial/Unknown | 1 | 1 | 2 | 2 | 6
  Non-Hispanic White | 506 | 498 | 482 | 520 | 2006
Region of Enrollment [Number; unit: participants]
  United States | 571 | 553 | 551 | 587 | 2262
Global Cognitive Composite [Mean (Standard Deviation); unit: z-scores] — The global composite is average of z-scores for each component. Each component has mean 0 at baseline, thus the composite z-score has mean 0. Individual component tests are 1) Telephone Interview for Cognitive Status-modified that measures global cognitive function, 2) Immediate and Delayed Story Recall tests for verbal memory, 3) Oral Trail Making Test for attention and executive function, 4) Verbal Fluency, 5) Number Span Test for attention and working memory, and 5) Digit Ordering Test for working memory. Higher positive scores reflect better performance. There are no clinical thresholds.
  z-scores | -0.01 (0.99) | 0.02 (1.00) | 0.05 (1.02) | -0.05 (0.99) | 0.00 (1.00)

OUTCOME MEASURES:

1. Primary Outcome: Global Cognitive Function: Average Change Over Follow-up From Baseline
Description: A composite cognitive measure that averages individual test z-scores of the Telephone Interview for Cognitive Status-modified (TICSm) Total and Long, the Immediate and Delayed Story Recall tests, the Oral Trail Making A and B tests (log-transformed), the Category Fluency and Verbal Fluency tests, and the Number Span Backward and Forward tests. Scores are ordered so that better performance corresponds to higher positive scores. Longitudinal data are used to create a linear contrast for the primary analysis to compare the difference between the average of scores at Years 1, 2, and 3 and the baseline score, i.e. (z1+z2+z3)/3 - z0, where z's denote the composited measures at baseline and years 1-3. This contrast is fitted using a random effects model for repeated measures. The primary comparison is for the margins of the factorial design: active cocoa flavonal (with or without active multivitamin) versus placebo flavonal (with or without active multivitamin).
Time Frame: From Baseline through Year 3
Population: Intention to treat -- All enrolled participants
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Cocoa Extract + Multivitamin: 2 capsules containing 500 mg/d cocoa extract; daily MTV
Arm/Group | Cocoa Extract + Multivitamin | Cocoa Extract + Multivitamin Placebo | Cocoa Extract Placebo + Multivitamin | Cocoa Extract Placebo + Multivitamin Placebo
Number analyzed (Participants) | 571 | 553 | 551 | 587
score on a scale | 0.24 (0.02) | 0.15 (0.02) | 0.20 (0.02) | 0.15 (0.02)
Statistical Analysis 1: Comparison: Cocoa Extract + Multivitamin vs Cocoa Extract + Multivitamin Placebo vs Cocoa Extract Placebo + Multivitamin vs Cocoa Extract Placebo + Multivitamin Placebo; Marginal comparisons from a repeated measures model using a linear contrast to estimate the mean differences between baseline versus average values across follow-up; Test type: Other — two-tailed test of the null hypothesis of no differences between groups; p < 0.05, Mixed Models Analysis — Not adjusted; Mean from linear contrast = 0.03, 95% CI 2-sided [-0.02 to 0.08], Standard Error of Mean 0.02 — Marginal effect of cocoa flavonal versus cocoa placebo based on the mean difference between linear contrasts; Wald test of a linear contrast from the mixed effects analysis....see protocol

2. Secondary Outcome: Composite Cognitive Function
Description: A composite cognitive measure that averages individual test z-scores of the Telephone Interview for Cognitive Status-modified (TICSm) Total and Long, the Immediate and Delayed Story Recall tests, the Oral Trail Making A and B tests (log-transformed), the Category Fluency and Verbal Fluency tests, and the Number Span Backward and Forward tests. Scores are ordered so that better performance corresponds to higher positive scores. Longitudinal data are used to create a linear contrast for the primary analysis to compare the difference between the average of scores at Years 1, 2, and 3 and the baseline score, i.e. (z1+z2+z3)/3 - z0, where z's denote the composited measures at baseline and years 1-3. This contrast is fitted using a random effects model for repeated measures. The comparison for this secondary outcome is based on the margins of the factorial design to compare multivitamin (with or without cocoa flavonal) with multivitamin placebo (with or without cocoa flavonal)
Time Frame: From baseline through year 3
Population: Complete randomized cohort
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cocoa Extract + Multivitamin | Cocoa Extract + Multivitamin Placebo | Cocoa Extract Placebo + Multivitamin | Cocoa Extract Placebo + Multivitamin Placebo
Number analyzed (Participants) | 571 | 553 | 551 | 587
score on a scale | 0.24 (0.02) | 0.15 (0.02) | 0.20 (0.02) | 0.15 (0.02)
Statistical Analysis 1: Comparison: Cocoa Extract + Multivitamin vs Cocoa Extract + Multivitamin Placebo vs Cocoa Extract Placebo + Multivitamin vs Cocoa Extract Placebo + Multivitamin Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — two-tailed test of the null hypothesis of no differences between groups; p < 0.05, Wald test — Not adjusted; Mean difference of linear contrasts = 0.07, 95% CI 2-sided [0.02 to 0.12], Standard Error of Mean 0.02 — Marginal effects of multivitamin versus multivitamin placebo; Wald test of a linear contrast from the mixed effects analysis....see protocol

3. Secondary Outcome: Incident Mild Cognitive Impairment
Description: Mild cognitive impairment based on centralized adjudication of cognitive test scores and input from a proxy. Limited to participants free of mild cognitive impairment at baseline. Incidence over 3 years of follow-up.
Time Frame: From baseline through year 3
Population: Limited to participants free of mild cognitive impairment at baseline. In a factorial design such as this, primary comparisons are cocoa flavanol vs cocoa flavanol placebo (pooling across multivitamin and multivitamin placebo) and multivitamin vs multivitamin placebo (pooling across cocoa flavanol and cocoa flavanol placebo). To provide outcomes for the four cells does not conform with the protocol or the published results and will not be consistent with the statistical analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Cocoa Extract: Daily cocoa extract (capsule containing 750 mg/d flavanols, including 75 mg (-)-epicatechin, and 90 mg theobromine)
- Cocoa Extract Placebo: Daily cocoa extract placebo
Arm/Group | Cocoa Extract | Cocoa Extract Placebo
Number analyzed (Participants) | 916 | 940
Participants | 47 | 63
Statistical Analysis 1: Comparison: Cocoa Extract vs Cocoa Extract Placebo; Test type: Equivalence — Proportional hazards regression -- unadjusted two-sided test; p = 0.15, Regression, Cox — Not adjusted; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.52 to 1.11] — Comparison group is placebo

4. Secondary Outcome: Incidence of Mild Cognitive Impairment Among Those Free at Baseline
Description: Mild cognitive impairment based on central adjudication of test scores with input from proxies. Based on test scores administered annually across 3 years.
Time Frame: From baseline through year 3
Population: Participants free of mild cognitive impairment at baseline. In a factorial design such as this, primary comparisons are cocoa flavanol vs cocoa flavanol placebo (pooling across multivitamin and multivitamin placebo) and multivitamin vs multivitamin placebo (pooling across cocoa flavanol and cocoa flavanol placebo). To provide outcomes for the four cells does not conform with the protocol or the published results and will not be consistent with the statistical analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Multivitamin: Daily multivitamin
- Multivitamin Placebo: Daily multivitamin placebo
Arm/Group | Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 920 | 936
Participants | 53 | 57
Statistical Analysis 1: Comparison: Multivitamin vs Multivitamin Placebo; Test type: Equivalence — Unadjusted 2-sided test; p = 0.62, Regression, Cox — Unadjusted; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.63 to 1.32] — Comparison group is placebo

5. Secondary Outcome: Executive Function
Description: Average of z-scores for the following tests: Oral Trail Making Test - B (log-transformed), Category Verbal Fluency, Letter Verbal Fluency, Number Span Test (Backwards and Forward). Higher (positive) scores reflect better performance. Linear contrast of scores collected at baseline, year 1, year 2, and year 3: (z1+z2+z3)/3 - z0)
Time Frame: From baseline through year 3
Population: All randomized participants. In a factorial design such as this, primary comparisons are cocoa flavanol vs cocoa flavanol placebo (pooling across multivitamin and multivitamin placebo) and multivitamin vs multivitamin placebo (pooling across cocoa flavanol and cocoa flavanol placebo). To provide outcomes for the four cells does not conform with the protocol or the published results and will not be consistent with the statistical analysis plan.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cocoa Extract | Cocoa Extract Placebo
Number analyzed (Participants) | 1144 | 1138
score on a scale | 0.06 (0.02) | 0.04 (0.02)
Statistical Analysis 1: Comparison: Cocoa Extract vs Cocoa Extract Placebo; Test type: Equivalence — Cocoa Flavonal minus Placebo; p = 0.24, Mixed Models Analysis — Unadjusted; Wald test comparing linear contrasts; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.02 to 0.08], Standard Error of Mean 0.03 — Cocoa Flavonal minus placebo

6. Secondary Outcome: Episodic Memory
Description: Average z-scores from Telephone Interview for Cognitive Status-modified Delayed Word List, Story Immediate Recall, Story Delayed Recall. Higher (positive) scores reflect better performance. Annual test administrations.
Time Frame: From baseline through year 3
Population: In a factorial design such as this, primary comparisons are cocoa flavanol vs cocoa flavanol placebo (pooling across multivitamin and multivitamin placebo) and multivitamin vs multivitamin placebo (pooling across cocoa flavanol and cocoa flavanol placebo). To provide outcomes for the four cells does not conform with the protocol or the published results and will not be consistent with the statistical analysis plan.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cocoa Extract | Cocoa Extract Placebo
Number analyzed (Participants) | 1144 | 1138
score on a scale | 0.29 (0.02) | 0.27 (0.02)
Statistical Analysis 1: Comparison: Cocoa Extract vs Cocoa Extract Placebo; Unadjusted 2-tailed test; Test type: Equivalence — two-sided; p = 0.41, Mixed Models Analysis — Unadjusted; Comparison of linear contrasts: cocoa flavonal minus placebo; Median Difference (Final Values) = 0.03, 95% CI 2-sided [-0.04 to 0.09], Standard Error of Mean 0.03 — Cocoa flavonal minus placebo

7. Secondary Outcome: Executive Function
Description: Average of z-scores for the following tests: Oral Trail Making Test - B (log-transformed), Category Verbal Fluency, Letter Verbal Fluency, Number Span Test (Backwards and Forward). Higher (positive) scores reflect better performance. Tests administered annually.
Time Frame: From baseline through year 3
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 1128 | 1140
score on a scale | 0.08 (0.02) | 0.02 (0.02)
Statistical Analysis 1: Comparison: Multivitamin; 2-sided test, unadjusted; Test type: Equivalence — 2 sided test, multivitamin minus placebo; p = 0.02, Mixed Models Analysis — Unadjusted; Comparison of linear contrasts; Mean Difference (Net) = 0.06, 95% CI 2-sided [0.01 to 0.11], Standard Error of Mean 0.03 — Multivitamin minus placebo

8. Secondary Outcome: Episodic Memory
Description: Average z-scores from Telephone Interview for Cognitive Status-modified Delayed Word List, Story Immediate Recall, Story Delayed Recall. Higher (positive) scores reflect better performance.
Time Frame: From baseline through year 3
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Multivitamin | Multivitamin Placebo
Number analyzed (Participants) | 1128 | 1140
score on a scale | 0.31 (0.02) | 0.25 (0.02)
Statistical Analysis 1: Comparison: Multivitamin vs Multivitamin Placebo; Multivitamin minus placebo; Test type: Equivalence — 2-sided, unadjusted; p = 0.04, Mixed Models Analysis — Unadjusted; Comparison of linear contrasts; Mean Difference (Net) = 0.06, 95% CI 2-sided [0.002 to 0.126], Standard Error of Mean 0.03 — Multivitamin minus placebo

ADVERSE EVENTS:
Time Frame: Across all follow-up -- 3 years.
Description: Mortality was collected by the parent trial and passed on to us. Adverse events were collected and published by the parent COSMOS trial, but were not separately passed on to us. Per instructions from the reviewer, because mortality was not collected by COSMOS-Mind, we now do not report it in this document.
Arm/Group | Cocoa Extract + Multivitamin | Cocoa Extract + Multivitamin Placebo | Cocoa Extract Placebo + Multivitamin | Cocoa Extract Placebo + Multivitamin Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03035201/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT03035201/SAP_001.pdf